CLINICAL TRIAL: NCT02688608
Title: Phase II Trial of Pembrolizumab in Metastatic or Locally Advanced Anaplastic/ Undifferentiated Thyroid Cancer
Brief Title: Pembrolizumab in Anaplastic/Undifferentiated Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Saad A Khan (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Saad A Khan, Assistant Professor of Medicine (Oncology), Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 012016-019; STU 012016-019 (Other: University of Texas Southwestern Medical Center)
Record Dates: First submitted 2016-01-20; First posted 2016-02-23 (Estimated); Results first posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Anaplastic Thyroid Cancer
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pembrolizumab (Experimental): 200 milligrams of Pembrolizumab will be given intravenously every 3 weeks.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg IV once every 3 weeks
  Other Names: Keytruda-Merck

SUMMARY:
This study is being done because there are currently no approved and no commonly working targeted therapies in anaplastic thyroid cancer (ATC). This is an area of urgent need for patients, not just for approved treatments but also rationally-designed clinical trials designed specifically for ATC. Patients diagnosed with anaplastic thyroid cancer have a very high likelihood of dying because of their disease. As such there is a clear need for improving therapy for ATC.

DETAILED DESCRIPTION:
The goal of this multi-center, open-label trial is to measure the impact of treating metastatic anaplastic thyroid cancer patients with immune checkpoint therapy. This trial will potentially lead to the development of new therapy for anaplastic thyroid cancer. The drug to be administered, pembrolizumab is FDA approved with known side effects and is active in many tumor types.

Programmed death 1 or (PD-1) PD-1/PD-L1 expression will be measured and reported for patients undergoing therapy with pembrolizumab. This will help determine if there PD-1 or PD-L1 are predictive biomarkers for anti-PD-1 therapy. It will also add to the data regarding their frequency in aggressive thyroid cancer. Where available, genomic profiling data will be analyzed to determine if there is a correlation between response and mutational status.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Histologically or cytologically confirmed diagnosis of anaplastic thyroid cancer or undifferentiated thyroid cancer. A diagnosis of possible ATC/UTC will be allowed if the clinical presentation is consistent with anaplastic or undifferentiated thyroid cancer.
3. Be ≥ 18 years of age on day of signing informed consent.
4. Have measurable disease based on RECIST 1.1.
5. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived sample.
6. Have a performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
7. Demonstrate adequate organ function as defined in the protocol. ,
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
10. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis).
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
18. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-10; Primary Completion 2020-10 (Actual); Study Completion 2021-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saad Khan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 6
Completed | 5
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (OR)
Description: Overall response (OR) represents those participants that collectively achieve either complete response (CR) or partial response (PR) within 18 months, as defined below per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
  * Complete Response (CR) = Disappearance of all target lesions
  * Partial Response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Overall Response (OR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s)
  * Stable disease (SD) = Small changes that do not meet any of the above criteria The outcome is reported as the cumulative number of participants receiving at least one dose of study treatment, that achieve either a CR or PR with 6 months, a number without dispersion.
Time Frame: up to 18 months.
Population: Response assessment data was not obtained for all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 5
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 3
  Overall Response (OR) | 3
  Stable disease (SD) | 1
  Progressive disease (PD) | 1

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) means to remain alive without disease progression. Progressive disease is defined as a 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s). The outcome is reported as the number of participants who received at least one dose of study treatment and remained alive without progression at 2 years after the beginning of treatment, a number without dispersion.
Time Frame: 2 years
Population: Survival data was not available for all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 5
Participants | 0

3. Secondary Outcome: Adverse Events Associated With Pembrolizumab
Description: Safety of the study treatment pembrolizumab is based on the number of adverse effects caused by pembrolizumab, referred to as related adverse events or toxicities. Reported adverse events (related) will be serious as defined by the Code of Federal Regulations at 21CFR§312.32, or non-serious. The outcome is reported as the number of non-serious and serious adverse events that occurred with the nominal study period (35 cycles or 2 years) that were reported as possibly, probably, or definitely related to pembrolizumab, a number without dispersion.
Time Frame: 2 years
Measure: Number; unit: related adverse events
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 6
related adverse events
  Non-serious Adverse Events | 35
  Serious Adverse Events | 1

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) means to remain alive without consideration of treatment response status.
  The outcome is reported as the number of participants who received at least one dose of study treatment and were known to remain alive at 2 years after the beginning of treatment, a number without dispersion. Subjects who become lost-to-follow-up before the 2-year assessment are not included.
Time Frame: 2 years
Population: Survival data was not available for all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events including grade 5 adverse events (death) are only reported for the adverse event collection period (2 years). Only adverse events and deaths occurring within 2 years are reported as adverse events.
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 5/6
Serious Adverse Events (participants affected / at risk) | 6/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Mucositis, oral (Gastrointestinal disorders) | 2 (2)
Neoplasm, other - disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Pain (General disorders) | 1 (1)
Parietal mass, right front (Nervous system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia, aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (General disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin irritation, pain at GI tube site (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=6)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Hypocalcemia (Blood and lymphatic system disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
Double vision (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1)
Intermittent Abdominal pain (Gastrointestinal disorders) | 1 (1)
Loss of sensation, lip (Gastrointestinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Oral Lesions (Gastrointestinal disorders) | 1 (1)
Pruritus (itching), lips (Gastrointestinal disorders) | 1 (1)
Trouble swallowing (Gastrointestinal disorders) | 4 (4)
Appetite change (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Cold intolerance (General disorders) | 1 (1)
Fatigue (General disorders) | 6 (15)
Focal weakness (General disorders) | 1 (1)
General Weakness (General disorders) | 1 (1)
Leg swelling (General disorders) | 3 (3)
Pain (General disorders) | 1 (1)
Redness (General disorders) | 2 (2)
Oral Lesions (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 3 (3)
ALK phosphate increase (Investigations) | 1 (1)
ALT/AST increase (Investigations) | 1 (1)
Elevated creatinine (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 2 (2)
Weight loss (Investigations) | 1 (1)
Diaphoresis (excessive sweating) (Metabolism and nutrition disorders) | 2 (2)
Arthritis (joint inflamation) (Musculoskeletal and connective tissue disorders) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
General Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, low back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, neck (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Sensory Change (Nervous system disorders) | 3 (3)
Speech change (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Polydipsia (Renal and urinary disorders) | 3 (3)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cough, dry (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough, productive (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough, wet (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (nosebleed) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intermittent cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seasonal allergies (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Shortness of breath, recumbent (orthopnea) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sputum production (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (itching) (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (itching), dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 6 (18)
Orthopnea (Vascular disorders) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT02688608/Prot_SAP_000.pdf